CLINICAL TRIAL: NCT00005575
Title: Psychophysiological Interactions in Non-Cardiac Chest Pain
Brief Title: Treatment of Non-Cardiac Chest Pain With Imipramine or Cognitive-Behavioral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: NCCP (completed); 42428-06
Record Dates: First submitted 2000-05-01; First posted 2000-05-02 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Chest Pain
Keywords: Imipramine; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Chest Pain | interventions — Imipramine; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Imipramine
Behavioral: Cognitive-behavior therapy

SUMMARY:
Approximately 75,000-150,000 patients each year in the United States undergo intensive cardiac evaluations for symptoms of angina-like chest pain that produce no positive findings. These patients often have high levels of disability and suffering and account for $250,000,000-$500,000,000 in estimated health care costs each year. There is some evidence from randomized, controlled trials that a pharmacologic agent, imipramine, and a program of training in pain coping skills and cognitive-behavioral therapy (CBT) both produce short-term reductions in pain intensity. However, no studies have compared the effects of these two treatments on measures of pain, suffering, and disability at post-treatment and over a one-year follow-up period.

Our investigation is a 16-week, randomized controlled outcome study of these interventions and their respective placebo control procedures. One hundred and sixty patients are being recruited for this study. We will assess the effects of our interventions on patients' pain levels, quality of life, and health care resource usage at baseline, post-treatment, 6-month follow-up, and at 12-month follow-up. We will evaluate the clinical significance of our treatment effects as well as their statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Substernal chest pain at least 2X per week for at least 3 months;
* Angiographic evidence of normal or non-obstructive (<50% luminal diameter narrowing) coronary arteries among subjects > 40 years of age; OR Normal exercise stress tests, normal echocardiogram, and cardiologist evaluation that symptoms are not cardiac in origin among subjects < 40 years of age;
* Gastroesophageal reflux disease ruled out by 24-hour pH monitoring, endoscopy, or 1-month trial of anti-reflux therapy with omeprazole 20 mg bid;
* Pain threshold levels for esophageal balloon distention must be 12 ml.

Exclusion Criteria:

* Mitral valve prolapse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Laurence A. Bradley, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Bradley LA, Richter JE, Scarinci IC, Haile JM, Schan CA. Psychosocial and psychophysical assessments of patients with unexplained chest pain. Am J Med. 1992 May 27;92(5A):65S-73S. doi: 10.1016/0002-9343(92)80059-9. PMID 1595768
- [Background] Mayou RA, Bryant BM, Sanders D, Bass C, Klimes I, Forfar C. A controlled trial of cognitive behavioural therapy for non-cardiac chest pain. Psychol Med. 1997 Sep;27(5):1021-31. doi: 10.1017/s0033291797005254. PMID 9300508
- [Background] Cannon RO 3rd, Quyyumi AA, Mincemoyer R, Stine AM, Gracely RH, Smith WB, Geraci MF, Black BC, Uhde TW, Waclawiw MA, et al. Imipramine in patients with chest pain despite normal coronary angiograms. N Engl J Med. 1994 May 19;330(20):1411-7. doi: 10.1056/NEJM199405193302003. PMID 8159194